CLINICAL TRIAL: NCT04396925
Title: Point-of-care Ultrasonography in Norwegian General Practice and Self-perceived Use in Diagnostics - a Prospective Observational Study
Brief Title: Point-of-care Ultrasonography in Norwegian General Practice
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Mette Brekke, Professor Mette Brekke, University of Oslo
Other Study IDs: 521500-710890-413601
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Point-of-care Ultrasound; General Practice; Family Medicine; Diagnostics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Point-of care Ultrasonography — GPs using POCUS and how it affects clinical judgement

SUMMARY:
The scope of this study is to explore how general practitioners (GPs) use Point-of-Care Ultrasonography (POCUS) in Norway. Thirty GPs will register information each time they use POCUS during a three-month period. Acquired information include the purpose of the scan, which organ is scanned, frequencies of POCUS and changes in diagnosis, plan, and treatment after the scan.

This is a strict observational study without any intervention.

DETAILED DESCRIPTION:
The scope of this prospective, observational study is to explore how general practitioners (GPs) use Point-of-care Ultrasonography (POCUS) in their daily practice and whether or not POCUS affects the diagnostic process. A similar study has previously by the university of Aalborg, Denmark with Clinical Trials ID NCT03375333. A part of this project is to assess the external validity of their questionaire.

POCUS use will be explored through reports of indication, frequency, consumed time both in total and the the scan, changes in diagnosis and further follow-up by the following questions:

What is the purpose of the planned scan? Which organ(s) do the GPs plan to scan? What is(are) the tentative diagnosis(-es) that warrants the use of POCUS? How would the GP follow-up the patient, if scanning was not possible? Would treatment be initiated? What kind of treatment?

The GP will register the precise time before and after the scan to assess how much time the use of POCUS adds to the consultation. The time spent scanning will also be registered to explore how much time is spent undressing/dressing the patient and booting the ultrasound device.

Which organ(s) was(were) scanned? How often are the GPs able to display the relevant structure(s) with POCUS? How confident are the GPs in their assessments? Did the scan alter the tentative diagnosis? What are the new diagnosis(es)? Did the scan alter the plan for further examination(s)? Did the scan alter the plan for further treatment?

The effect on the diagnostic process will be investigated through the reported change(s) in the tentative diagnosis after the use of POCUS. The GPs' confidence in the scans will also be evaluated. The aims are to describe:

Do POCUS change the GPs' tentative diagnosis? Do POCUS increase the confidence of the GPs' tentative diagnosis? What is the relationship between the experience of GPs' confidence and the change in the tentative diagnoses? Is there a relationship between change from symptom diagnoses to disease diagnoses? What was the relationship between scanned organs and the GPs' confidence in the tentative diagnosis? What was the effect on the treatment of patients?

This will be explored through changes in the planned follow-up or need for further treatment for the patient. The aims are to describe:

Did POCUS change the GPs' plan for further examinations of the patient Did POCUS change the planned treatment for the patient

Study setting:

Norwegian day-time general practice

Interventions:

This study do not involve any new interventions. The GPs involved in this study already use POCUS as at part of their clinical practices.

Sample size Norway has approximately 4700 GPs. A recent study states that 30% of Norwegian GPs used POCUS in 2016. Most of these GPs scans less than one monthly. Duration of registration is three months. Of the entire GP population, 30 GPs will be included in this study. If the participating GPs scan twice weekly on average, the aim is to achieve 720 scans.

Recruitment

Participating GPs:

GPs using POCUS will be recruited through the continuous post-graduate small-group education, ultrasonography networks, participation in conferences, through teaching sessions, and through contacts via the Norwegian association for ultrasonography in general practice.

Participating patients:

No direct patient data will be used, only the assumed diagnosis and changes to these.

There are no restrictions made regarding age or gender.

Base-line assessment of GPs The will not be an assessment of the GPs' skills in the use of POCUS. Any GP is allowed to scan regardless of formal skills

Data collection A questionnaire is made for both electronic and manual registration. SurveyXact is the online database used for electronic registration. The questionnaire includes a time log to ensure the before and after registration. Several pilot tests have been and will be performed both in the research group and with GPs using POCUS to ensure comprehension, feasibility and compliance.

The GPs will be asked to access a questionnaire in SurveyXact each time they use their ultrasound device during their daily work. The GPs can access the questionnaire via mobile phone, iPad or computer, using a unique link (respondent link) allocated each participating GP. A key file, connecting each participating GP with the respondent link in SurveyXact (link), will be safely stored at the Research Unit for General Practice in Aalborg.

Questions before scanning are the following:

GP ID number What is the main reason to use POCUS in this patient? (Rule-in/Rule-out, Explore, Scan a known condition, Screening or Other) Which organs/positions is expected to be scanned? (organs on list) What is the main tentative diagnosis for this patient? (ICPC2 codes) Are there any other possible tentative diagnoses in this case? (ICPC2 codes) What is the overall plan for this patient? (Acute admission to hospital, Subacute referral to hospital, Elective referral hospital, Subacute referral to specialist, Elective referral to specialist, Referral to radiology, Other referral e.g. physiotherapist, Follow-up in the clinic, No plan for follow-up, Other) Which treatment will be initiated at this stage? (medical treatment, referral for treatment, initiated other treatment, None, Other)

Questions after the performed scanned:

Time used on the POCUS examination? (minutes) Which organs/positions were scanned? (organs on list) Was the GP able to produce ultrasound images of the relevant structures of (inserted text) ? (yes, no - please specify) What did the GP find? (Certain positive findings, Uncertain positive findings, Certain negative findings, Uncertain negative findings, Incidental findings - please specify in free text) Before POCUS the following tentative diagnoses were registered (inserted text) Has this changed? (yes but the ICPC-2 code is unchanged, Yes both diagnosis and ICPC-2 code have changed, no) What is the tentative diagnosis for this patient now? (ICPC-2 codes) Are there any other possible tentative diagnoses for this patient (please specify)? (ICPC-2 codes) How is the GPs confidence in their main tentative diagnosis, after POCUS? (Highly increased confidence, More confident, unchanged confidence, Less confident, Highly reduced confidence) Before POCUS the following plan was registered (inserted text) for the patient. Has this plan changed? (yes, no) What is the overall plan for this patient, now? (Acute admission to hospital, Subacute referral to hospital, Elective referral hospital, Subacute referral to specialist, Elective referral to specialist, Referral to radiology, Other referral e.g. physiotherapist, Follow-up in the clinic, No plan for follow-up, Other) Before POCUS the following treatment was registered (inserted text) for the patient. Has the treatment changed? (yes, no) Which treatment will be initiated at this stage? (medical treatment, referral for treatment, initiated other treatment, None, Other)

Statistics The data will be analyzed using descriptive statistics. Multivariate regression analysis will be used to analyze whether traits of the GP affect the results of the scans.

Research ethics approval

The study has an approval from the Norwegian Center for Research Data.

As this study is an observational study, and does not include any intervention, approval by the Norwegian Regional Committee for medical and Health Research Ethics was granted.

Protocol amendments will be declared and all editions. Any changes to the protocol will be saved.

ELIGIBILITY:
Inclusion Criteria:

General practitioners who use point-of-care ultrasound in day time general practice

Exclusion Criteria:

* Conflict of interest, e.g. if the GP is part of the research group or if the GP has direct financial interest in selling US devices.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners who use point-of-care ultrasonography as a part of clinical practice. Out-of-hours scanning excluded
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
How general practitioners use POCUS in their daily practice | 2024
  The GPs' indications for the use of point-of-care ultrasound (POCUS) will be described through the number and type of scans performed, and through frequencies of the tentative diagnoses that warrant the use of POCUS. The frequency of each POCUS examination (numerator) will be compared to all performed scans (denominator). The GPs will register the time used for the POCUS examination. By the before and after registration of the organs intended to scan and the organ actually scanned, the extent of modification of tentative diagnosis, plan for further examination and/or treatment.

SECONDARY OUTCOMES:
How GPs evaluate their confidence | 2024
  The GPs state a tentative diagnosis as one main and other possible diagnoses before the use of POCUS. After the scan, the GPs will see their tentative diagnosis prior to the scan. The GPs are asked if these diagnoses have changed. Has the diagnosis changed, they will be asked to specify this. The tentative diagnosis is registered as ICPC-2 codes. The GPs assess their confidence in the tentative diagnoses after the use of POCUS: Increased confidence, more confident, unchanged confidence, less confident, reduced confidence. To test the reliability of the GPs' declaration of confidence, we examine if an increased confidence is correlated to specific organs scanned (Q2.2), a reduction in the total number of diagnoses (Q1.3, Q1.4, Q2.6 and Q2.7), or a change from symptom diagnosis to disease diagnosis.
Characteristics of the physician that influence the effect of POCUS | 2024
  The effect on changes in tentative diagnoses, diagnostic confidence and plan for patients including treatment. We aim to describe:
  * Does the gender of the GP affect any of these outcomes?
  * Do the years of clinical experience affect any of these changes?
  * Do the years of POCUS experience affect any of these changes?
  * Are there geographical variations in the performed scans?

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brekke, Professor, Study Chair — University of Oslo, Department of General Practice; Hans-Christian Myklestul, M.D., Principal Investigator — University of Oslo, Department of General Practice; Trygve Skonnord, PhD, Study Director — University of Oslo, Department of General Practice
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data registered are available for the cooperating researchers at the university in Aalborg Denmark. The purpose of further analyses is to compare the external validity of the questionnaire.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2025
Access Criteria: The data are only available for cooperating researchers in Aalborg, Denmark including Martin Bach Jensen and Camilla Aakjaer Andersen

REFERENCES:
- [Result] Aakjaer Andersen C, Brodersen J, Davidsen AS, Graumann O, Jensen MBB. Use and impact of point-of-care ultrasonography in general practice: a prospective observational study. BMJ Open. 2020 Sep 17;10(9):e037664. doi: 10.1136/bmjopen-2020-037664. PMID 32948563
- See also: URL to the study published in BMJ Open — https://bmjopen.bmj.com/content/10/9/e037664